CLINICAL TRIAL: NCT01168375
Title: The Role of Umbilical Cord Serum Therapy on Improvement of Corneal Epithelial Defect Following Diabetic Vitrectomy
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Collaborators: Ophthalmic Research Center (Ambiguous)
Responsible Party: Ophthalmic Research Center
Other Study IDs: 8742
Record Dates: First submitted 2010-07-01; First posted 2010-07-23 (Estimated); Last update posted 2010-07-23 (Estimated); Status verified 2010-03

CONDITIONS: Corneal Epithelial Defect

ARMS (2):
- conventional therapy (Active Comparator): chloramphenicol and betamethasone eye drops every 6 hours, cycloplegic (homatropine) eye drop every 8 hours
  Interventions: Drug: conventional therapy
- conventional therapy plus umbilical cord serum eye drop (Active Comparator)
  Interventions: Drug: conventional therapy plus umbilical cord serum eye drop

INTERVENTIONS:
Drug: conventional therapy plus umbilical cord serum eye drop — chloramphenicol and betamethasone eye drops every 6 hours, cycloplegic (homatropine) eye drop every 8 hours plus umbilical cord serum eye drop 20% every 4 hours
  Arms: conventional therapy plus umbilical cord serum eye drop
Drug: conventional therapy — chloramphenicol and betamethasone eye drops every 6 hours, cycloplegic (homatropine) eye drop every 8 hours
  Arms: conventional therapy

SUMMARY:
80 diabetic patients underwent vitrectomy and had no history of Eye herpes infection, Refractive surgery, Autoimmune disease, Immune deficiency will be randomized into two groups (double blind)to evaluate the role of umbilical cord serum therapy on improvement of corneal epithelial defect following diabetic vitrectomy. Both groups will take the conventional medication including Chloramphenicol, Betamethasone, Cycloplegic eye drops besides the case group will take umbilical cord serum eye drop in the eye operated. After surgery the corneal epithelial defect will be measured by slit lamp.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic patients with corneal epithelial defect following diabetic vitrectomy at labbafinejad Hospital

Exclusion Criteria:

* Any history of Eye herpes infection, Refractive surgery, Autoimmune disease, Immune deficiency
* Patients with one eye
* Use of any eye drops except Chloramphenicol, Betamethasone, Cycloplegic and contact lens for corneal epithelial defect

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

PRIMARY OUTCOMES:
measurement of corneal epithelial defect
  measurement of corneal epithelial defect in days 3,5,7,12 by slit lamp

CONTACTS AND LOCATIONS:
Locations (1):
- Ophthalmic Research Center, Tehran, Tehran Province, Iran